CLINICAL TRIAL: NCT02954081
Title: Real-world Benefit of Apremilast Treatment of Patients With Moderate-to-severe Psoriasis After Transition From Fumaric Acid Esters
Brief Title: APremilast After FumaRic Acid Ester Treatment
Acronym: APART
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-10004-PSOR-024
Record Dates: First submitted 2016-11-01; First posted 2016-11-03 (Estimated); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Phase I: Fumaric acid esters. Phase II: Apremilast — Apremilast

SUMMARY:
Patient treatment preference and treatment satisfaction of physicians and patients comparing fumaric acid ester therapy with subsequent apremilast treatment

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 years
* Moderate to severe plaque-type psoriasis according to SmPC
* Phase I: Patients will be included once they are started on systemic fumaric acid esters (e.g. Fumaderm initial®) for the treatment of moderate-to-severe psoriasis vulgaris. Patients initiated on fumaric acid esters will be followed for a maximum of 24 weeks during phase I. Patients continued on fumaric acid esters beyond 24 weeks or switched to a therapy other than apremilast during or at the end of the 24-week phase I period will no longer be followed.
* Phase II: Patients switched to apremilast during or at the end of the 24-week phase I period will be included in phase II and followed for additional 32 weeks.
* Written informed consent

Exclusion Criteria:

* Prior treatment with biologics
* According to SmPC
* Participation in another clinical trial (parallel inclusion in the National psoriasis registry PsoBest is allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Adult patients ≥18 years
  * Moderate to severe plaque-type psoriasis according to SmPC
Sampling Method: Probability Sample
Enrollment: 687 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Mean absolute value of the overall TSQM score at week 24 of apremilast (APR) therapy (phase II). | 56 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Site, Hamburg, Germany

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Expanded Access for CC-10004 — https://clinicaltrials.gov/ct2/show/NCT02954081?term=CC-10004-PSOR-024&rank=1